CLINICAL TRIAL: NCT00273845
Title: Reducing Barriers to Drug Abuse Treatment Services
Acronym: RBP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wright State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Marianne Shreck, Wright State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-407-10; 1R01DA015690 (NIH); HSP 2527
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Substance Abuse
Keywords: case management; substance abuse treatment; linkage
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): One session of motivational interviewing
  Interventions: Behavioral: Motivational interviewing
- 2 (Experimental): Five sessions of strengths-based case management
  Interventions: Behavioral: Strengths-Based Case Management

INTERVENTIONS:
Behavioral: Motivational interviewing — One session
  Arms: 1
Behavioral: Strengths-Based Case Management — 5 sessions
  Arms: 2

SUMMARY:
The broad goal of this study is to assess the effectiveness of two interventions to facilitate treatment linkage and treatment engagement. "Treatment linkage" is operationally defined as completion of agency intake procedures and attendance at the first clinical or therapy session. "Treatment engagement" represents a more comprehensive conceptualization of "treatment retention" and includes measures of the clinical and ancillary services actually received by the client over time; as such, client engagement focuses on the intensity and duration of treatment participation. This study will enhance the CIU concept by conducting a controlled trial, using a three-armed research design, of interventions designed to enhance treatment linkage and treatment engagement. These interventions - a Motivational Intervention and Strengths-Based Case Management - are science-based and have demonstrated efficacy in moving drug abusers towards treatment and supporting treatment engagement.

DETAILED DESCRIPTION:
The Specific Aims of the project are:

1. To conduct a detailed qualitative/ethnographic investigation to study: (a) the processes and factors operant in a person's decision to link with a substance abuse treatment agency once a formal (i.e., professional) assessment and referral have been made; and (b) the processes and factors operant in staying in treatment once it has been initiated.
2. To identify and classify, using quantitative methods, the operant barriers to treatment linkage and engagement. We will assess the factors that are associated with these barriers and examine the effects of the study's interventions on removing them.
3. To evaluate the effectiveness, using a controlled trial, of a Motivational Intervention and Strengths-Based Case Management, compared to the CIU's "standard" referral process, by examining differences between the Standard, Motivational Intervention, and Case Management conditions on treatment linkage and engagement outcomes. The conceptual framework for this controlled trial is the well-studied Andersen model of access and health service use, modified for chemical dependency services (Andersen, 1995). The interventions are designed to affect mutable factors such as perceived barriers to treatment. Data will be collected at baseline, and at 3 and 6 months thereafter. Analyses will examine whether the interventions work better with different groups of clients (e.g. cocaine users versus marijuana users, males versus females, different ethnicities, etc); as well as different treatment modalities (standard outpatient versus intensive outpatient.)
4. To conduct a quantitative investigation of the effects of Individual Level and Health Care System Level factors that predict treatment linkage and engagement in the context of the proposed interventions. This study component will develop comprehensive models to predict how these factors interact with the study's interventions to effect treatment linkage and treatment engagement.

ELIGIBILITY:
Inclusion Criteria:

* substance abuse or dependence per DSM-IVR criteria

Exclusion Criteria:

* active thought disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2003-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Linkage and Retention in substance abuse treatment | 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Rapp, M.S.W., Principal Investigator — Boonshoft School of Medicine, Wright State University
Locations (1):
- Samaritan CrisisCare, Dayton, Ohio, United States